CLINICAL TRIAL: NCT02579876
Title: A Double, Blind Placebo-controlled, Randomized Trial to Study Efficacy and Safety of the Viaskin Milk for Treating Milk Induced Eosinophilic Esophagitis in Children
Brief Title: Milk Patch for Eosinophilic Esophagitis
Acronym: SMILEE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: DBV Technologies (Industry)
Responsible Party: Principal Investigator, Antonella Cianferoni, Assistant Professor, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-010148
Record Dates: First submitted 2015-10-14; First posted 2015-10-20 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Eosinophilic Esophagitis; Milk Allergy
Keywords: Milk Allergy; Viaskin Milk; Epicutaneous ImmunoTherapy (EPIT); Eosinophilic Esophagitis; Milk-Induced Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis; Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Viaskin Milk 500 mcg (Active Comparator): Viaskin patch containing milk protein. The patch is applied to the skin
  Interventions: Drug: Viaskin Milk 500 mcg
- Viaskin Placebo (Placebo Comparator): Viaksin patch without any milk protein.
  Interventions: Drug: Viaskin Placebo

INTERVENTIONS:
Drug: Viaskin Milk 500 mcg — Biological: Viaskin Milk 500 mcg Subjects epicutaneously administered daily (up to 24 hours application per day) with a patch containing 500 mcg cow's milk proteins.
  Other Names: Milk Patch; Viaskin Epicutaneous ImmunoTherapy (EPIT)
  Arms: Viaskin Milk 500 mcg
Drug: Viaskin Placebo — Biological: Viaskin Placebo Subjects epicutaneously administered daily (up to 24 hours application per day) with a patch containing a matching placebo formulation.
  Other Names: Placebo Patch; Placebo Epicutaneous ImmunoTherapy (EPIT)
  Arms: Viaskin Placebo

SUMMARY:
This is a single-site, double-blind, placebo-controlled, randomized trial to study efficacy and safety of the Viaskin® Milk Patch for children with milk induced Eosinophilic Esophagitis (EoE). 20 subjects will be randomized 3:1 to Viaskin® Milk or placebo patch.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized trial to study the efficacy and safety of Viaskin® Milk, an allergen extract of milk administered epicutaneously using the Viaskin® epicutaneous delivery system (EPIT) in subjects from 4 to 17 years old with a milk induced Eosinophilic Esophagitis. Subjects will be randomized in a 3:1 ratio into two different treatment groups, to receive EPIT with Viaskin® Milk (500 µg of milk proteins) or placebo.

Subjects who complete the double-blind treatment period (approximately 11 months), will automatically rollover into an open label treatment period (additional 11 months). All subjects will receive the 500 µg (micrograms) Viaskin Milk patch.

ELIGIBILITY:
Inclusion Criteria:

* Well-documented medical history of Eosinophilic Esophagitis after ingestion of milk and currently following a strict milk-free diet.
* Upper endoscopy and biopsy at initial clinical evaluation during Visit 2 showing greater than 15 eosinophils/high power field (HPF) isolated to the esophagus meeting the consensus diagnosis of Eosinophilic Esophagitis, after milk was re-introduced into the subject's diet (30 ml/day for 1 week to 2 months), while the subject was on proton pump inhibitor.
* Upper endoscopy and biopsy at second clinical evaluation during Visit 3 showing less than 5 eosinophils per HPF isolated to the esophagus after a minimum of 6 weeks under milk-free diet, and while the subject is on proton pump inhibitor.
* Negative pregnancy test for female subjects of childbearing potential. Females of childbearing potential must use effective method of contraception to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of participation in the study. Sexual abstinence will be accepted as an effective method of contraception for girls below 18 years of age.
* Subjects and/or parents/guardians willing to comply with all study requirements during their participation in the study.
* Signed informed consent from parent(s)/guardian(s) of children < 18 years + children's assent.
* Subjects agree to maintain a constant diet during the trial, with the exception of milk.
* Subjects will maintain constant medications for asthma and allergic rhinitis during the trial.

Exclusion Criteria:

* Subjects with a history of severe anaphylaxis to milk with the following symptoms: hypotension, hypoxia, neurological compromise (collapse, loss of consciousness or incontinence), Quincke Edema or requiring intubation.
* Active IgE- mediated milk allergy.
* Pregnancy or lactation.
* Subjects with other eosinophilic gastrointestinal disorders.
* Subjects on swallowed corticosteroids or anti-leukotrienes for Eosinophilic Esophagitis.
* Subjects with symptomatic allergy to pollens whose symptoms during the corresponding pollen season might interfere with the recording of symptoms during the upper endoscopy/biopsy, if the upper endoscopy/biopsy is conducted during the pollen season. The Investigator will have to ensure that the period for conducting the upper endoscopy for such a subject will be outside of the pollen season.
* Subjects treated with systemic long-acting corticosteroids (depot corticosteroids) within 12 weeks prior to Visit 1 and/or systemic short-acting corticosteroid within 4 weeks prior to Visit 1 or any systemic corticosteroid at screening.
* Subjects with asthma conditions defined as follows:

  1. Uncontrolled persistent asthma by National Asthma Education and Prevention Program Asthma guidelines (2007).
  2. at least two systemic corticosteroid courses for asthma in the past year or one oral corticosteroid course for asthma in the past three months;
  3. prior intubation for asthma in the past two years.
* Subjects on β-blocking agents, angiotensin-converting enzyme inhibitors, angiotensin receptor blockers, calcium channel blockers or tricyclic antidepressant therapy.
* Subjects undergoing any type of immunotherapy to any food within one year prior to Visit 1.
* Subjects presently on aeroallergen immunotherapy and unwilling or unable to discontinue.
* Subjects currently treated with anti-tumor necrosis factor drugs or anti-Immunoglobulin E (IgE) drugs or any biologic immunomodulatory therapy within one year prior to Visit 1.
* Allergy or known hypersensitivity to placebo excipients either of the Viaskin® or Tegaderm®.
* Subjects suffering from generalized dermatologic diseases with no intact skin zones to apply the Viaskin®, or urticarial and mast cell disorders such as chronic idiopathic urticaria.
* Subjects (or parents of subjects) with obvious excessive anxiety and unlikely to cope with the conditions of an upper endoscopy and biopsy.
* Past or current disease(s), which in the opinion the sponsor-investigator, may affect the subject's participation in this study including but not limited to active autoimmune disorders, immunodeficiency, malignancy, uncontrolled diseases (hypertension, psychiatric (especially anxiety), cardiac), or other disorders (e.g., liver, gastrointestinal, kidney, cardiovascular, pulmonary disease, or blood disorders).
* Any history of drug or alcohol abuse in the past five years.
* Subjects unable to follow the protocol and the protocol requirements.
* Participation in another clinical intervention study in the three months prior to Study Visit 1.
* Subjects on any experimental drugs or treatments.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12-20 (Actual); Study Completion 2018-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Cianferoni, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spergel JM, Elci OU, Muir AB, Liacouras CA, Wilkins BJ, Burke D, Lewis MO, Brown-Whitehorn T, Cianferoni A. Efficacy of Epicutaneous Immunotherapy in Children With Milk-Induced Eosinophilic Esophagitis. Clin Gastroenterol Hepatol. 2020 Feb;18(2):328-336.e7. doi: 10.1016/j.cgh.2019.05.014. Epub 2019 May 14. PMID 31100455

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Viaskin Milk 500 mcg | Viaskin Placebo
Started | 15 | 5
Completed | 14 | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Viaskin Milk 500 mcg | Viaskin Placebo | Total
Number analyzed (Participants) | 15 | 5 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 5 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.46 (2.99) | 12.71 (2.03) | 10.69 (3.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 10 | 5 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 5 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 5 | 20
Eosinophils (Eos) per high power field (HPF) on Milk [Mean (Standard Deviation); unit: Eos/hpf] | 72.4 (29.52) | 60.93 (49.39) | 64 (44.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum Esophageal Eosinophil Count From Baseline to End of Double-blind Treatment. (Intent to Treat Population)
Description: Esophageal biopsy samples will be obtained prior to randomization and after completion of treatment. Intraepithelial eosinophils will be counted in all high powered fields (HPFs) using light microscopy. A HPF will be counted only if at least half of the field is occupied by tissue. The maximum eosinophil count per HPF will be reported for each esophageal biopsy site (at each of 2 levels).
  The maximum eosinophil count for each patient will be calculated from either level. For the final outcome, mean from each individual patients maximum eosinophil count/hpf along with standard deviation will be calculated.
Time Frame: From baseline to month 11 (end of double blind phase)
Measure: Mean (Standard Deviation); unit: Eosinophils (Eos)/high power field (HPF)
Arm/Group | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 14 | 5
Eosinophils (Eos)/high power field (HPF) | -10.8 (37.73) | -24.2 (63)

2. Primary Outcome: Change in Eosinophils/High Power Field at End of Double-blind (DB) (Per Protocol Patients)
Description: as for outcome 1
Time Frame: Month 11(end of double blind phase)
Measure: Mean (Standard Deviation); unit: Eosinophils (Eos)/high power field
Arm/Group | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 7 | 2
Eosinophils (Eos)/high power field | -26.86 (22.53) | 42.5 (31.82)

3. Secondary Outcome: Eosinophilic Esophagitis Symptom Score (Intent to Treat Population)
Description: Symptoms of Eosinophilic Esophagitis range from abdominal pain, gastroesophageal reflux, vomiting, and difficult swallowing. Investigator assessment of the subject's symptoms was completed on a 4-point Likert scale for 3 separate symptoms (vomiting, abdominal pain and dysphagia).
  Investigator assessment of the subject's symptoms was completed on a 4-point Likert scale for 3 separate symptoms (vomiting, abdominal pain and dysphagia). (0-none, 1-mild, 2-moderate, 3-severe, ). Total score is reported with a range of 0 to 9. A lower score is better.
Time Frame: Total Symptom Score at End of DB Phase, Month 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 14 | 5
units on a scale | 1.07 (1.49) | 1.40 (1.14)

4. Secondary Outcome: Esophageal Endoscopy Score (ITT)
Description: Upper endoscopies with biopsies (2 each of proximal and distal, plus any inflamed areas) will be completed before and after each treatment period. Each endoscopy will be scored using a validated standardized measure which examines 4 major esophageal features (rings, furrows, exudates and edema) and the presence of minor features of narrow caliber esophagus, feline esophagus, stricture and crepe paper esophagus. Each feature is graded: 0-none, 1 mild, 2-moderate, 3-severe. The scores are summed including both minor and major criteria.
  Total score is presented and lower score is better. The range is from 0-12
Time Frame: At end of DB phase, at 11 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 14 | 5
score on a scale | 1.93 (1.58) | 1.60 (1.67)

5. Secondary Outcome: Eosinophils Per HPF at End of Double Bind Protocol (Per Protocol) Patients
Description: Maximum Eosinophils/HPF after milk reintroduction at the end of double bind phase
Time Frame: End of DB Phase, at 11 months
Measure: Mean (Standard Deviation); unit: Eos/hpf
Arm/Group | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 7 | 2
Eos/hpf | 25.57 (31.19) | 95 (63.64)

6. Secondary Outcome: Pediatric Eosinophilic Esophagitis Symptom Score (ITT)
Description: Measure of Pediatric Eosinophilic Esophagitis symptom Score (PEESS) at the end of DB phase for the Intent to Treat Population The PEESS® is a 20 question survey asking patient symptom intensity and frequency on a 5 point scale (0 to 4) for each question for the preceding month. Therefore, the total score can range from 0 to 80. The total score is reported and lower score is better
Time Frame: Month 11, end of Double Blind Phase
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 14 | 5
units on a scale | 11.15 (11.07) | 13.2 (7.33)

7. Secondary Outcome: Endoscopy Score (Per Protocol Patients)
Description: Upper endoscopies with biopsies (2 each of proximal and distal, plus any inflamed areas) will be completed before and after each treatment period. Each endoscopy will be scored using a validated standardized measure which examines 4 major esophageal features (rings, furrows, exudates and edema) and the presence of minor features of narrow caliber esophagus, feline esophagus, stricture and crepe paper esophagus. Each feature is graded: 0-none, 1 mild, 2-moderate, 3-severe. The scores including both major and minor criteria are summed.
  Total score is presented and lower score is better. The range is from 0-12
Time Frame: Month 11 (end of double blind phase)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 7 | 2
score on a scale | 1.43 (1.51) | 3 (1.41)

8. Secondary Outcome: Pediatric Eosinophil Esophagitis Symptom Score (PP Population)
Description: Pediatric Eosinophilic Esophagitis Symptom Score at end of DB phase using the validated Pediatric Eosinophilic Esophagitis Symptom Score (PEESS).The PEESS® is a 20 question survey asking patient symptom intensity and frequency on a 5 point scale (0 to 4) for each question for the preceding month. Therefore, the total score can range from 0 to 80. The total score is reported and lower score is better.
Time Frame: Month 11, End of Double Blind Placebo Control
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 7 | 2
score on a scale | 12.2 (8.57) | 17 (1.41)

ADVERSE EVENTS:
Time Frame: The length of time is 1 year from the start of the study to end of double blind phase
Description: All adverse events (AEs) were collected from the start of the study. . All Treatment emergent AEs are reported
Arm/Group | Viaskin Milk 500 mcg | Viaskin Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/5
Other Adverse Events (participants affected / at risk) | 15/15 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viaskin Milk 500 mcg (N=15) | Viaskin Placebo (N=5)
Vocal Cord Dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viaskin Milk 500 mcg (N=15) | Viaskin Placebo (N=5)
General GI Symptoms (Gastrointestinal disorders) | 10 (10) | 2 (2)
Upper Respiratory Infections (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Administration Site Conditions (General disorders) | 12 (12) | 5 (5)
Ear infections (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Muscloskeletal (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Infections (Infections and infestations) | 8 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT02579876/SAP_000.pdf
  • Study Protocol (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT02579876/Prot_001.pdf